CLINICAL TRIAL: NCT04958382
Title: A Single Center, Randomized, Single Blind, Exploratory Study for Evaluating the Efficacy of Ciprofol in Patients Under Narcotic Sleep With Chronic Insomnia
Brief Title: Study for Evaluating the Efficacy of Ciprofol in Patients Under Narcotic Sleep With Chronic Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Mengchang Yang, Deputy Chief Physician, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK3486-IIT-01
Record Dates: First submitted 2021-06-24; First posted 2021-07-12 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol (Experimental)
  Interventions: Drug: ciprofol
- placebo (Placebo Comparator)
  Interventions: Drug: medium/long chain fat emulsion injection (C8-24Ve)

INTERVENTIONS:
Drug: ciprofol — intravenous infusion of ciprofol at 0.12 mg/kg, followed by 0.4-1.6 mg/kg/h for maintenance
  Arms: Ciprofol
Drug: medium/long chain fat emulsion injection (C8-24Ve) — at the infusion rate of 25-30 mL/h
  Arms: placebo

SUMMARY:
This is a single center, randomized, single blind, exploratory clinical study.About 30 patients with chronic insomnia are planned to be enrolled in this study and randomized into two groups by a ratio of 4:1 (Figure 1), with group 1 (24 subjects) for ciprofol and group 2 (6 subjects) for placebo (fat emulsion). Cognitive behavioral therapy (CBT) will be given to these patients during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 (inclusive) to 70 (inclusive) years old;
2. ASA class of I-II;
3. With chronic insomnia refractory to conventional drugs in the past 3 months (benzodiazepine receptor agonists and other drugs). Other drugs: melatonin, melatonin receptor agonists, and traditional Chinese medicine;
4. Compliant with the diagnostic criteria of ICSD-3 chronic insomnia:

   1. At least one of the following chief complaints: initial insomnia, difficulty in sleep maintenance, early awakening, refusal to go to bed at an appropriate time, and difficulty in falling asleep without nursing;
   2. At least one of the following daytime symptoms: tiredness, short tempered, work/study/social skills decreased;
   3. Occurrence of the above symptoms at least 3 times per week and lasting for more than 3 months;
5. Voluntarily adopt narcotic sleep and obtain the written informed consent form.

Exclusion Criteria:

1. With contraindications to deep sedation/general anesthesia or a history of past sedation/anesthesia accidents;
2. With a history of allergy or contraindications to anesthetics;
3. With a medical history or evidence of any of the followings before screening/at baseline, which may increase sedation/anesthesia risks:

   1. History of cardiovascular diseases: uncontrolled hypertension [systolic blood pressure (SBP) ≥ 170 mmHg and/or diastolic blood pressure (DBP) ≥ 105 mmHg without treatment, or SBP > 160 mmHg and/or DBP > 100 mmHg despite antihypertensive treatment], severe arrhythmia, heart failure, Adams-stokes syndrome, New York Heart Association (NYHA) Class ≥ III, severe superior vena cava syndrome, pericardial effusion, acute myocardial ischemia, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medical treatment, II-III degree atrioventricular block (excluding patients with pacemakers);
   2. History of respiratory system disorders: respiratory insufficiency, history of obstructive pulmonary disease, history of bronchospasm requiring treatment within 3 months before screening, and acute respiratory tract infection with obvious symptoms such as fever, wheezing, nasal obstruction, and cough within 1 week before baseline;
   3. History of neurological and psychiatric disorders: craniocerebral injury, possible convulsions, myoclonus, intracranial hypertension, cerebral aneurysms, history of cerebrovascular accidents; schizophrenia, mania, insanity, history of cognitive disorder; history of epilepsy; mental disorder suggested by Mini International Neuropsychiatric Interview (MINI);
   4. History of gastrointestinal disorders: gastrointestinal retention, active hemorrhage, or conditions that may lead to reflux and aspiration;
   5. History of blood donation or blood loss of ≥ 400 mL within 3 months before screening;
4. With the following airway management risks at screening:

   1. History of asthma or stridor;
   2. Sleep apnea syndrome;
   3. History or family history of malignant hyperthermia;
   4. History of tracheal intubation failure;
   5. Judged by investigators to have difficult airway or judged as difficult tracheal intubation (modified Mallampati class IV) at screening;
5. Receipt of any of the following medications/therapies at screening/baseline:

   1. Any clinical study within 1 month before screening;
   2. Sedatives/anesthetics, and/or sedative-hypnotics within 72 h before baseline;
   3. Antidepressants and anxiolytics within 14 days before baseline;
6. Laboratory test abnormalities at screening:

   1. Total bilirubin > 2 × ULN (upper limit of normal);
   2. Aspartate aminotransferase (AST) and alanine transaminase (ALT) > 2 × ULN;
   3. Blood creatinine > 1.5 × ULN;
7. Unable to fast for 6 h before dose administration;
8. With a history of smoking, drug abuse and/or positive urine drug screening results, or positive breath alcohol test results at baseline and/or a history of alcohol abuse within 3 months before screening. Alcohol abuse is defined as an average of > 2 units of alcohol consumed per day (1 unit = 360 mL of beer with 5% alcohol, 45 mL of liquor with 40% alcohol, or 150 mL of wine);
9. Pregnant or breastfeeding females; women of child-bearing potential or men who are unwilling to use contraception during the trial; or patients who are planning pregnancy within 1 month after the trial (including male patients);
10. Unable to avoid engaging in dangerous occupations requiring concentration and/or motor coordination 72 h after administration;
11. Judged by investigators to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Polysomnography (PSG) | Day -2 to Day 90
  total sleep time (TST)
Polysomnography (PSG) | Day -2 to Day 90
  sleep latency (SL)
Polysomnography (PSG) | Day -2 to Day 90
  wake after sleep onset (WASO)
Sleep log | Day -2 to Day 90
  subjective total sleep time (sTST)
Sleep log | Day -2 to Day 90
  subjective sleep-onset latency (sSOL)
Sleep log | Day -2 to Day 90
  subjective wake after sleep onset (sWASO)

SECONDARY OUTCOMES:
Self-rating scales | Day -2 to Day 90
  Pittsburgh Sleep Quality Index (PSQI)（0-21）
Self-rating scales | Day -2 to Day 90
  Insomnia Severity Index (ISI)（0-28）
Self-rating scales | Day -2 to Day 90
  PHQ-9 Depression Test Questionnaire（0-27）
Self-rating scales | Day -2 to Day 90
  GAD-7 Anxiety Test Questionnaire（0-21）
Self-rating scales | Day -2 to Day 90
  Epworth Somnolence Scale（0-24）;

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Sichuan, China